CLINICAL TRIAL: NCT02865395
Title: Timing of B and O Suppositories to Help Relieve Post-operative Bladder Spasms and Urinary Discomfort in Patients Undergoing Lithotripsy
Brief Title: Timing of B and O Suppositories to Help Relieve Post-operative Bladder Spasms
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Another study published with similar results
Sponsor: Campbell Grant (Other)
Responsible Party: Sponsor-Investigator, Campbell Grant, Urology Resident, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GW051534
Record Dates: First submitted 2016-02-17; First posted 2016-08-12 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Overactive Bladder
Keywords: Belladonna and Opium Suppositories
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pre-operative Suppository (Experimental): A B&O Suppository will be placed in the patient's rectum after the induction of anesthesia, but before the surgery.
  Interventions: Drug: Belladonna and Opium Suppository
- Post-operative Suppository (Active Comparator): A B&O Suppository will be placed in the patient's rectum while still under anesthesia, but after the surgery.
  Interventions: Drug: Belladonna and Opium Suppository
- Rectal Exam (Placebo Comparator): Patient's will be given a rectal exam after the procedure but while still under anesthesia to serve as a placebo.
  Interventions: Procedure: Rectal Exam

INTERVENTIONS:
Drug: Belladonna and Opium Suppository
  Arms: Post-operative Suppository; Pre-operative Suppository
Procedure: Rectal Exam
  Arms: Rectal Exam

SUMMARY:
Ureteroscopy is a common procedure in Urology that patients undergo daily to deal with a variety of ailments. These procedures often require that the bladder be filled and emptied with sterile water or saline several times during the procedure, and often result in the patient receiving a catheter at the end of the procedure. One common side effect is that patients experience bladder spasm or discomfort for a period of time after these procedures. Belladonna and Opium (B and O) suppositories and PO Oxybutynin are often given in the post-operative setting to relieve these symptoms.

The principle objectives of this study are:

1. To determine if the addition of a B and O supprette suppository at the end of cystoscopic/ureteroscopic procedures reduces the incidence of bladder spasms and urinary discomfort that patients experience in the post-operative setting.
2. To determine if using peri-operative B and O supprette suppositories reduces the need for pos-operative oral Ditropan and use of narcotic pain medications.

DETAILED DESCRIPTION:
The patients will be divided into three research arms. Patients will be randomly selected for one of the groups using a random number generator between 1 and 3. There will be a "Control Group" which will receive a rectal exam while still in the operating room in the lithotomy position after the procedure. There will be a "Postoperative OR" group which will receive a B and O suppository while still in the operating room in the lithotomy position after the procedure. Finally, there will be a "Preoperative OR" group which will receive a B and O suppository after the induction of anesthesia prior to beginning the urologic procedure in the lithotomy position. The "Control Group" will receive a rectal exam in the operating room after the procedure but before extubation to simulate the effects of suppository administration so that the investigators know that any effects are due to the medication and not to the placement of the suppository itself. Those patients in the "control group" may receive a B and O suppository as part of standard procedure in the post-operative period if these individuals experience any bladder spasms and wish to have this as a treatment. This administration will be at the discretion of the operating surgeon as it is in standard cases. Patients may also receive Ditropan in the post-operative setting, which is part of the standard procedure for treating bladder spasms following urologic procedures. Patients in the postoperative and preoperative OR groups will be offered Ditropan for any bladder spasms in the post-operative setting to control symptoms, which is part of the normal standard of care for anyone who has already received a B and O suppository with inadequate control of symptoms. All patients will be treated with a normal post-operative pain regimen which may include narcotics. This will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lithotripsy procedure at GW Hospital

Exclusion Criteria:

* The criteria for exclusion for those patients who agree to participate in the study will be patients with glaucoma, severe hepatic or renal disease, bronchial asthma, respiratory depression at the time of administration, convulsive disorders, allergy to anti-muscarinics or opiates, history of anorectal surgery, pre-operative use of antimuscarinics, chronic pain, chronic use of analgesics, or a history of alcohol or opioid dependency.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mufarrij, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-operative Suppository: A B&O Suppository will be placed in the patient's rectum after the induction of anesthesia, but before the surgery.
  Belladonna and Opium Suppository
- Post-operative Suppository: A B&O Suppository will be placed in the patient's rectum while still under anesthesia, but after the surgery.
  Belladonna and Opium Suppository
- Rectal Exam: Patient's will be given a rectal exam after the procedure but while still under anesthesia to serve as a placebo.
  Rectal Exam
Period: Overall Study
Arm/Group | Pre-operative Suppository | Post-operative Suppository | Rectal Exam
Started | 6 | 10 | 7
Completed | 0 (Data Not Collected) | 0 (Data Not Collected) | 0 (Data Not Collected)
Not Completed | 6 | 10 | 7
Not completed — Physician Decision | 6 | 10 | 7

BASELINE CHARACTERISTICS:
Population: We did not collect the data on any of these patients. Therefore there is no data on ethnicity, age, or sex.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-operative Suppository | Post-operative Suppository | Rectal Exam | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Participants

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Morphine Equivalent Dose
Description: No results collected on the post-operative morphine equivalent dose
Time Frame: 24 hours
Population: Study terminated prior to results.
Arm/Group | Pre-operative Suppository | Post-operative Suppository | Rectal Exam
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Post-Operative Pain
Description: Patients will be asked to fill out a short questionnaire with the faces scale to grade their pain on a scale of 1-10
Time Frame: 24 hours
Population: Data was not collected on these patients.
Arm/Group | Pre-operative Suppository | Post-operative Suppository | Rectal Exam
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Data collected over 2 months while study was recruiting patients. No adverse events recorded.
Description: No adverse events were reported.
Arm/Group | Pre-operative Suppository | Post-operative Suppository | Rectal Exam
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT02865395/Prot_SAP_000.pdf